CLINICAL TRIAL: NCT07332273
Title: Effect of Levothyroxine as Adjuvant Therapy to a Hypocaloric Diet in the Treatment of Obesity: a Randomized Placebo-controlled Trial.
Brief Title: Levothyroxine as Adjuvant to a Hypocaloric Diet for the Treatment of Obesity.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LEVOBESITY
Record Dates: First submitted 2025-09-05; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Thyroxine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Levothyroxine 88mcg (Experimental)
  Interventions: Drug: Levothyroxine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levothyroxine — Film-coated oral tablets containing levothyroxine 88 mcg, taken once daily for 9 months. All participants receive a structured lifestyle program: months 0-3 hypocaloric Mediterranean diet (~600 kcal/day deficit) with physical-activity advice; months 3-9 normocaloric Mediterranean diet with continued advice. The IMP is purchased from authorized manufacturers, then reconditioned and relabeled per GMP and supplied blinded for the full study period. Dispensing follows the randomization code; emergency unblinding only via the hospital pharmacy. Store per label (do not store above 25 °C); adherence assessed by pill count and self-report.
  Arms: Levothyroxine 88mcg
Drug: Placebo — (white, plain, circular), oral once daily for 9 months, no active ingredient. Administered alongside the same lifestyle program as the active arm (months 0-3 hypocaloric Mediterranean diet; months 3-9 normocaloric Mediterranean diet). Placebo is reconditioned and relabeled per GMP to be indistinguishable from levothyroxine; supply is blinded and dispensed per randomization code. Emergency unblinding is performed only by the pharmacy service when medically necessary.
  Arms: Placebo

SUMMARY:
Obesity is a chronic disease with high relapse rates after initial weight loss. Thyroid hormones modulate energy expenditure, body composition, and thermogenesis; higher TSH within the reference range and subclinical hypothyroidism have been associated with adverse metabolic profiles and weight gain. These signals suggest the thyroid axis could influence weight-loss response and subsequent regain. Levothyroxine (LT4) is widely used for hypothyroidism; evaluating its adjuvant role in obesity management is clinically relevant.

This is a phase III, randomized, double-blind, placebo-controlled, multicentre clinical trial conducted in five Spanish hospitals. A total of 286 adults (25-60 years) with grade I-II obesity will be enrolled if they have subclinical hypothyroidism (TSH 5-10 mIU/L with normal peripheral hormones) or are euthyroid with TSH in the highest tertile of the reference range. Participants are randomized 1:1, stratified by age, sex, and BMI.

Intervention: LT4 88 µg once daily or matching placebo for 9 months. During months 0-3, all participants receive a structured hypocaloric Mediterranean diet (≈600 kcal/day deficit; macronutrients 45% carbohydrates, 35% fats, 20% proteins) plus standardized physical-activity advice. From months 3-9, lifestyle support continues with a normocaloric Mediterranean diet. Physical-activity guidance targets ≥150 min/week of moderate-to-vigorous activity (spread over ≥3 days) and 2-3 resistance sessions/week.

Primary endpoint (3 months): change in body weight (kg and %) and body composition (BMI, waist/hip circumferences, fat mass, fat-free mass, total body water by bioimpedance) comparing LT4 versus placebo under the same lifestyle program. The study is powered for n=286.

Key secondary endpoints (up to 9 months): prevention of weight regain; changes in obesity stage; cardiometabolic markers (lipids, glucose/HbA1c, HOMA-IR, adipokines, inflammation, blood-pressure patterns); resting energy expenditure by indirect calorimetry; objectively measured physical activity by accelerometry; cardiac parameters (ECG) and safety; quality of life (EuroQol-5D). Mechanistic substudies assess adipose-tissue metabolic activity (gene/protein expression, browning markers, mitochondrial DNA) and explore gut microbiota, epigenetic signatures, nitrogen balance, and sex-specific differences in response.

Assessments are performed at baseline and follow-up visits through 9 months and include anthropometry, bioimpedance, laboratory panels, indirect calorimetry, ambulatory blood-pressure monitoring, ECG, diet/physical-activity questionnaires, and biobanking of blood, urine, and stool; an adipose-tissue biopsy is obtained in a subsample.

The trial uses intention-to-treat analyses with mixed linear models and is designed with 90% power to detect a clinically meaningful between-group difference in 3-month weight loss; total sample size is 286 (143 per arm). Overall study duration is 21 months (12 months of recruitment plus 9 months of treatment/follow-up); each participant remains in the study for 9 months.

In summary, this trial tests whether adding LT4 88 µg/day to a structured Mediterranean-diet and exercise program enhances early weight loss and helps prevent regain versus placebo in adults with obesity and high-normal TSH or subclinical hypothyroidism, while characterizing metabolic mechanisms and biomarkers of response.

ELIGIBILITY:
Inclusion Criteria:

* Adults 25-60 years of age.
* Obesity grade I-II: BMI 30.0-39.9 kg/m².
* Either subclinical hypothyroidism (TSH 5-10 mIU/L with normal peripheral hormones) or euthyroid with TSH in the highest tertile of the population reference range (no known thyroid disease).
* Able and willing to provide written informed consent.
* Women of childbearing potential: not pregnant or breastfeeding and using a highly effective contraception method (failure rate <1%) per CTCG guidance (e.g., hormonal methods, IUD/IUS, sterilization, or dual barrier with spermicide).

Exclusion Criteria:

* Diabetes mellitus (HbA1c ≥6.5%, fasting glucose ≥126 mg/dL, or 2-h OGTT ≥200 mg/dL).
* Any prior thyroid disease (hyperthyroidism, overt hypothyroidism) or prior LT4 treatment.
* Current or recent (≤3 months) use of levothyroxine, hypoglycaemic agents, antibiotics, or regular probiotics/prebiotics.
* Active cancer or cancer within the last 5 years (except basal-cell carcinoma).
* Chronic liver disease with total bilirubin ≥2.0 mg/dL or AST >3× ULN.
* Established cardiovascular disease (e.g., stroke, ischemic heart disease, peripheral artery disease).
* Atrial fibrillation or any arrhythmia history.
* Uncontrolled hypertension (>160/100 mmHg) despite therapy (assessed by ABPM at screening).
* Any heart failure; resting HR >85 bpm; eGFR <60 mL/min.
* Known HIV, HBV, or HCV infection.
* Acute inflammatory disease or inflammatory bowel disease.
* Serious underlying disease that, in the investigator's judgment, could affect participation.
* Drug/alcohol abuse, life expectancy <12 months, inability to follow the recommended diet or attend visits.
* Positive pregnancy test, pregnant, expecting pregnancy, or breastfeeding.
* Hypersensitivity to any component of the investigational product.
* Inability or unwillingness to provide informed consent.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 286 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Change in body weight (kg) from baseline to Month 3 | Baseline to Month 3 (12 weeks ±2)
Change in fat mass (kg) by bioimpedance from baseline to Month 3 | Baseline to Month 3 (12 weeks ±2)

SECONDARY OUTCOMES:
Weight-regain (kg) from Month 3 to Month 9 | Month 3 to Month 9 (36 weeks ±2)
Change in BMI (kg/m²) from baseline to Month 9 | Baseline to Month 9
Change in waist circumference (cm) from baseline to Month 9 | Baseline to Month 9
Change in fasting LDL-cholesterol (mg/dL) from baseline to Month 9 | Baseline to Month 9
Change in glycaemic control (HbA1c, %) from baseline to Month 9 | Baseline to Month 9
Change in insulin resistance (HOMA-IR) from baseline to Month 9 | Baseline to Month 9
Change in resting energy expenditure (kcal/day) by indirect calorimetry from baseline to Month 9 | Baseline to Month 9
Change in physical activity level measured by accelerometry | Baseline to Month 9
  Physical activity will be quantified by accelerometry using the ActiGraph WGT3X-BT device, worn for 7 consecutive days before and after the intervention periods, as specified in the protocol.
Change in blood pressure parameters assessed by ambulatory blood pressure monitoring (ABPM) from baseline to Month 9 | Baseline to Month 9
  Ambulatory blood pressure monitoring (24-hour ABPM) will be performed to register possible blood pressure adverse events, as specified in the protocol.
Change in heart rate measured by electrocardiogram (ECG) from baseline to Month 9 | Baseline to Month 9
  Cardiac evaluation will be performed by electrocardiogram (ECG). Minimum, maximum and average heart rates will be assessed as specified in the protocol.
Change in number of ventricular extrasystoles measured by electrocardiogram (ECG) from baseline to Month 9 | Baseline to Month 9
  The number of ventricular extrasystoles will be assessed by electrocardiogram (ECG) during cardiac evaluation, according to the protocol.
Change in QT interval measured by electrocardiogram (ECG) from baseline to Month 9 | Baseline to Month 9
  QT interval will be evaluated by electrocardiogram (ECG) as part of the cardiac assessment described in the protocol.
Incidence of adverse events (AEs) and serious adverse events (SAEs) | From first dose to Month 9
Change in quality of life measured by EuroQol-5D index from baseline to Month 9 | Baseline to Month 9
Change in quality of life measured by EuroQol-5D visual analogue scale (VAS) from baseline to Month 9 | Baseline to Month 9
Change in gene expression related to metabolic activity in adipose tissue (subsample) | Baseline to Month 3
  Gene expression changes in adipose tissue samples related to lipogenic and lipolytic capacity, adipokines, thyroid receptor and browning biomarkers will be analyzed, as described in the protocol.
Change in protein abundance related to metabolic activity in adipose tissue (subsample) | Baseline to Month 3
  Protein abundance changes in adipose tissue samples related to metabolic activity will be evaluated according to the protocol.
Change in mitochondrial DNA in adipose tissue (subsample) | Baseline to Month 3
  Mitochondrial DNA in adipose tissue samples will be analyzed as part of the metabolic activity assessment described in the protocol.
Change in gut microbiota diversity determined by 16S rRNA gene sequencing from baseline to Month 9 | Baseline to Month 9
Change in relative abundance of gut microbiota taxa determined by 16S rRNA gene sequencing from baseline to Month 9 | Baseline to Month 9
Change in nitrogen balance (g/day) from baseline to Month 9 | Baseline to Month 9

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Hospital Puerta del Mar, Cadiz
  - Hospital Reina Sofía, Córdoba
  - Hospital Universitario de Jaén, Jaén
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Clínico Universitario de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the published results and the data dictionary will be made available to the scientific community via institutional repositories, following FAIR principles and Spanish/EU data protection law (LOPD 3/2018; GDPR). Participants are informed about data use and re-use; personal identifiers are removed and study data are stored on encrypted, password-protected servers. Access will be provided after primary results publication, subject to a reasonable request and a data use agreement consistent with GDPR; supporting documents (protocol, SAP, blank CRFs) and code will also be shared.